CLINICAL TRIAL: NCT04377776
Title: Observational Study to Assess the Health Status of Transplanted Patients (Kidney or Pancreas or Pancreatic Islet Transplantation) at Transplant Medicine Unit (MITRA) During the COVID-19 Pandemic
Brief Title: Observational Study Concerning COVID-19 Infection in Transplanted Kidney, Pancreas or Pancreatic Islet Patients
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Antonio Secchi, Medicine Transplant Unit Director, IRCCS San Raffaele
Other Study IDs: COVID-19 MITRA
Record Dates: First submitted 2020-05-05; First posted 2020-05-06 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Kidney Transplant; Pancreas Tranplant; Pancreatic Islet Transplantation
Keywords: COVID-19 infection; Transplanted patients; kidney transplant; pancreas transplant; pancreatic islet transplantation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transplanted patients: Transplanted Kidney, Pancreas or Pancreatic Islet patients at MedicineTransplant Unit - San Raffaele Scientific Istitute
  Interventions: Other: Practice details

INTERVENTIONS:
Other: Practice details — Questionnaire

SUMMARY:
Collect informations on the health status of transplanted patients (kidney, kidney / pancreas, pancreas or pancreatic islet) during the COVID-19 pandemic. All informations will be collected by short questionnaire via phone.

ELIGIBILITY:
Inclusion Criteria:

Transplanted Kidney or Kidney/Pancreas or Pancreas or Pancreatic Islet patients at Transplant Medicine Unit - San Raffaele Scientif Institute

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transplanted Kidney, Pancreas or Pancreatic Islet patients
Sampling Method: Probability Sample
Enrollment: 644 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Global Prevalence of COVID-19 TX | From 01st February 2020 to 18 May 2020
  Global Prevalence of COVD-19 infection in transplanted patients
Hospitalization rate in COVID-19 TX | From 01st February 2020 to 18 May 2020
  Hospitalization rate of transplanted patients

SECONDARY OUTCOMES:
Correlation COVID-19 TX and type of transplantation | From 01st February 2020 to 18 May 2020
  Correlation between type of transplantation to COVID-19 virus infection
Prevalence of COVID-19 TX in italian provinces | From 01st February 2020 to 18 May 2020
  Prevalence COVID-19 virus infection in transplanted patients in italian provinces
Symptoms in COVID-19 TX | From 01st February 2020 to 18 May 2020
  Prevalence of different symptoms in COVID-19 virus infection in transplanted patients
Correlation COVID-19 TX and comorbidities | From 01st February 2020 to 18 May 2020
  Correlation between comorbidities to COVID-19 virus infection
COVID-19 TX Therapies | From 01st February 2020 to 18 May 2020
  Impact of different therapies on COVID-19 virus infection in transplanted patients
COVID-19 TX in family settings | From 01st February 2020 to 18 May 2020
  Impact of COVID-19 virus infection in transplanted patients family settings

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Secchi, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy